CLINICAL TRIAL: NCT03264833
Title: Accuracy and Precision Test of TempTraq® Compared to Pulmonary Artery Catheter for Monitoring Temperature in Adults in Intensive Care Unit
Brief Title: Accuracy and Precision Comparison of Temptraq
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Blue Spark Technologies (Unknown)
Responsible Party: Principal Investigator, Sandra Siedlecki, Senior Nurse Scientist, The Cleveland Clinic
Other Study IDs: NCT-03264833
Record Dates: First submitted 2017-02-02; First posted 2017-08-29 (Actual); Results first posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-01

CONDITIONS: Temperature

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: TempTraq — sensor-based external thermometer withmonitoring capability

SUMMARY:
Purpose The purpose of this feasibility study is to assess the accuracy and precision of the Temp-Traq thermometer for monitoring body temperature in adult patients under three conditions (hypothermia, normothermia, and hyperthermia).

Specific Aims

1. To assess the accuracy of the Temp-Traq thermometer as compared to a gold standard (Core temp measured by Pulmonary Artery Catheter)
2. To assess the precision of the Temp-Traq thermometer over repeated measures
3. To determine if accuracy &/or precision is consistent in three conditions (hypothermia, normothermia, or hyperthermia)

DETAILED DESCRIPTION:
Design A repeated measures within-group comparative design will be used for this study.

Sample/Setting To address the specific aims of this study the investigators will identify patients who have a pulmonary artery (PA) catheter in place (patients in intensive care units). Letters of support are attached from the unit managers where the study will take place (see attached).

Procedure Once a patient is identified, the researcher will record basic demographic data (see data collection form attached) and the axillary area will be assessed for visible signs of any skin conditions. If there are no visible signs of a skin condition the researcher will apply the Temp-Traq thermometer to the right or left axilla of the subject and record the location of the placement. The researcher will record both the PA and Temp-Traq recordings of subject's temperature (taken at the same time) on the data collection form (see attachment) at four data points; baseline (5 minutes post application of Temp-Traq) and every two hours (+/- 15 minutes) after baseline X 3. Previous testing of the TempTraq® on children and healthy adults has not resulted in any adverse skin reactions. However, as this is a new thermometer format and there is not a significant body of literature on potential skin reactions, the investigators will assess skin before and after application. Thus, at the end of the last reading the Temp-Traq thermometer will be removed and the skin will be assessed for erythema. If erythema is present the patient's nurse and physician will be notified by the researcher.

Protection of Human Subjects Since non-invasive temperature monitoring poses no risk to patients and is part of usual care and since the investigators will not collect or record any protected health information (PHI), written informed consent will not be sought. Patients will be identified by their study ID number only. The data will be collected by a registered nurse data collector familiar with the intensive care setting and data will be stored in a locked file cabinet in the researchers locked office. Temperature data for the Temp-Traq is collected through the Temp-Traq Application (AP) which will be placed on a Cleveland Clinic Approved and encrypted i-pad. Once the study is completed and all data has been transferred to the study database, the Temp-Traq application and all of its data will be deleted from the i-pad.

Analysis The investigators will use the TOST (Two One Sided t-tests) method for equivalence testing. This method requires a defined range of mean differences between two test methods, an estimate of the precision of the measurement of the two systems, and an estimate of the size of the possible difference in the means of the two methods under consideration. The TOST null hypothesis is a joint null hypothesis that the mean measurement differences between the two methods is greater than a critical lower bound and less than a critical upper bound. If the null is rejected then the investigators can conclude that the absolute difference of the means between Temp Traq and PA catheter falls within the specified range. It was determined that to be considered equivalent with respect to accuracy the mean measurements of the two methods should be within ± 0.2 degrees of each other. Precision tests for Temp-Traq thermometer using accepted ASTM test methods for various combinations of temperature and humidity provided a range of measurement variation between .0000435 and .019928 with a mean of 0.000254500. If the investigators assume both test methods exhibit the same levels of precision then the variance of the differences between their two means will reduce to two times the values listed previously. This will result in estimates of the standard deviations of the mean differences of .0093, .032, and .063 respectively.

The two methods for body temperature that will be examined are core temperature measurements with a PA catheter and temperature measurements using the Temp-Traq (measured in degree Celsius simultaneously). Paired temperature measurements for both methods will be taken simultaneously every 2 hours for a 6 hour period. This will provide 4 repeated temperature measures per patient. The simultaneous measurements within a given patient should exhibit a high degree of correlation. If .7 is chosen as the lower bound for the correlation between the paired readings (higher correlations would result in an estimate of fewer patient samples thus the choice of .7 is conservative) and if the average standard deviation of the mean of the differences is used as an estimate of the expected variability, then it would be possible to declare measurement equivalence for a difference of ±.19 with a sample size of 40 patients. This assumes the ASTM measurements of instrument variation are representative of the within patient variance. Given the vagaries of patient-to-patient this may be too optimistic an estimate.

A sample size of at least 40 patients will provide 80% or greater power for testing for equivalence between methods where the mean difference is .1 or less for up to a ten-fold increase in the estimates of the variability of the differences based on the ASTM precision measures and for a mean difference of .15 for up to a five-fold increase in these same measures. If the sample size is 40 then the power for the test of equivalence, where the difference is .15 and the standard deviation is a ten-fold increase, is 35%. Agreement testing: The Bland-Altman test will be used to test the agreement of the two methods. This test will permit a check for significance of bias between the two measures (the average difference between the two measures) as well as a check for significant trending over the range of the measurements. If the bias is significant then the results of the two differ by an overall offset in their measurements. If the trending (slope of the regression line) is significant then the difference between the two measurements changes as their magnitude changes which means the two methods are not in agreement.

The only measurements of instrument precision are those provided by the ASTM assessment. It is reasonable to assume the within patient measurement variation will be greater than the measurements from the controlled testing. A sample size of at least 40 patients is, from a statistical standpoint, a reasonable number and this sample size provides acceptable power for a mean difference of .1 for a ten-fold increase in the estimate of minimum test variability. This sample size will also provide enough data for the Bland-Altman test for agreement. Because this is a repeated measures test and even one missing measurement will impact the results, the investigators plan to over-sample in order to assure the study has the power to answer the questions posed.

ELIGIBILITY:
Inclusion Criteria:

Inclusion Criteria Adult patient (male or female) in intensive care unit who will have a PA catheter in place for at least the next 8 hours; and who have no visible skin condition to the axillary region upon inspection by the research nurse are eligible for this study

Exclusion Criteria:

1. Patients younger than 21
2. Patients who will not have a PA catheter in place for the next 8 hours
3. Patients who have a visible skin condition to the axillary region upon inspection by the research nurse
4. Patients who will be going for procedures or for some reason will not be available for the 6 hours of the study

Min Age: 21 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: To address the specific aims of this study the investigators will identify at least 40 patients who have a pulmonary artery (PA) catheter in place (patients in intensive care units).
Sampling Method: Non-Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2016-12-15 (Actual); Primary Completion 2017-09-01 (Actual); Study Completion 2017-10-01 (Actual)

IPD SHARING:
Plan to Share IPD: No
IPD will not be shared

REFERENCES:
- [Background] Eliades, A, Stoner, K. and Frisone, J. (unpublished paper) Use of skin patch device to obtain temperature measurements
- [Background] Farnell S, Maxwell L, Tan S, Rhodes A, Philips B. Temperature measurement: comparison of non-invasive methods used in adult critical care. J Clin Nurs. 2005 May;14(5):632-9. doi: 10.1111/j.1365-2702.2004.00916.x. PMID 15840078
- [Background] Lawson L, Bridges EJ, Ballou I, Eraker R, Greco S, Shively J, Sochulak V. Accuracy and precision of noninvasive temperature measurement in adult intensive care patients. Am J Crit Care. 2007 Sep;16(5):485-96. PMID 17724246
- [Background] Pinsky MR, Vincent JL. Let us use the pulmonary artery catheter correctly and only when we need it. Crit Care Med. 2005 May;33(5):1119-22. doi: 10.1097/01.ccm.0000163238.64905.56. PMID 15891346
- [Background] Sund-Levander M, Grodzinsky E. Assessment of body temperature measurement options. Br J Nurs. 2013 Aug 8-Sep 12;22(15):880, 882-8. No abstract available. PMID 24052967

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited in a medical ICU over a 6 month period
Groups:
- Longitudinal Single Arm Study: Patients were assessed at baseline, hour 2, hour 4 and hour 6 Temperature (Celsius) data were compared between TempTraq reading and pulmonary artery (central, internal; used as the gold standard) readings at 4 time points
Period: Overall Study
Arm/Group | Longitudinal Single Arm Study
Started | 60
Completed | 60
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Longitudinal Single Arm Study: Medical ICU patients with a pulmonary artery catheter; obtained core temp (PA catheter) and compared to TempTraq temperatures in Celsius
Arm/Group | Longitudinal Single Arm Study
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.8 (11.13)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 40
Race/Ethnicity, Customized [Number; unit: participants]
  White | 40
  Black | 20
pulmonary artery catheter core temperature sensor [Mean (Full Range); unit: Degree Celsius] — PA- (central venous catheter) body temperature in Celsius Temp Traq body temperature in Celsius
  Degree Celsius
    PA-Celsius | 36.84 [31.9 to 39]
    TempTraq- Celsius | 36.3 [31.9 to 39]

OUTCOME MEASURES:

1. Primary Outcome: Temperature Comparison
Description: Core temperature monitoring (degree Celsius) with temp-Traq thermometer compared to Pulmonary Artery (PA) catheter
Time Frame: Multiple time points up to 6 hours post thermometer placement
Population: Adults in a medical intensive care unit with pulmonary artery catheter monitoring that included core temperature
Measure: Mean (95% Confidence Interval); unit: Degree Celsius
Groups:
- Longitudinal Single Arm Study: Mean differences in Core temperature (degree Celsius) monitoring with temp-Traq thermometer compared to Pulmonary Artery (PA) catheter
Arm/Group | Longitudinal Single Arm Study
Number analyzed (Participants) | 60
Degree Celsius
  Initial placement | -0.60 [-0.78 to -0.42]
  2 hours post placement | -0.24 [-0.39 to -0.097]
  4 hours post placement | -0.16 [-0.30 to -0.03]
  6 hours post placement | -0.19 [-0.37 to -0.02]
  Cumulative change | -0.30 [-0.39 to -0.22]

ADVERSE EVENTS:
Time Frame: 6 hours
Description: No adverse events reported. (Patients were assessed for rash or erythema)
Arm/Group | Longitudinal Single Arm Study
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-07): https://cdn.clinicaltrials.gov/large-docs/33/NCT03264833/Prot_SAP_000.pdf